CLINICAL TRIAL: NCT00755144
Title: A Prospective Randomized Study on Early Clinical and Functional Outcome of the ROCC and LCS Total Knee Arthroplasty Implant Designs
Brief Title: A Randomized Control Trial to Assess Early Clinical and Functional Outcome of the ROCC and LCS Total Knee Implant Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMET UK 05
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): ROCC
  Interventions: Device: ROCC Knee
- 2 (Active Comparator): LCS
  Interventions: Device: LCS Knee

INTERVENTIONS:
Device: LCS Knee — Cementless total knee arthroplasty with LCS Knee
  Arms: 2
Device: ROCC Knee — Cementless total knee arthroplasty with ROCC Knee
  Arms: 1

SUMMARY:
This is a prospective Randomised Control Trial to compare the Early Clinical and Functional Outcome of the ROCC and LCS total knee arthroplasty implant designs.

DETAILED DESCRIPTION:
This study compares two similar designs of cementless rotating bearing total condylar knee replacements. The study will be conducted at a single clinical unit with a senior orthopaedic surgeon implanting all devices.Their performances will be assessed by clinical scores and comprehensive function outcome documentation undertaken by qualified physiotherapists. The persons undertaking the assessments will be blinded to which implants the patients have.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for cementless knee replacement
* Patients skeletally mature and under 80 years of age at pre-operative clinic
* Patients presenting with osteoarthritis of the knee
* Patients must be ambulatory at time of pre-operative clinic
* Patients must be able to understand instructions and be will to return for follow-up

Exclusion Criteria:

* Previous knee surgery (except arthroscopic/open menisectomy)
* Patients with inflammatory arthritis
* Patients with significant medical co-morbidity - ASA IV
* Disorders causing abnormal gait or significant pain
* Patients unable to consent
* Severe visual impairment

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
American Knee Society Score | Preoperative, 8weeks, 1 year

SECONDARY OUTCOMES:
WOMAC | preoperative, 8 weeks, 1 year
VAS Pain | Preoperative, 4weeks, 8weeks, 3months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Musgrave Park Hospital, Belfast, United Kingdom